CLINICAL TRIAL: NCT04788719
Title: Pre and Postoperative Gait Analysis of Randomized Patients to 2 Different Cement Fixation Methods
Brief Title: Pre and Postoperative Gait Analysis of Randomized Patient to 2 Different Cement Fixation Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Pre and post op gait analysis
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Gait Analysis; Hip Arthritis; Total Hip Arthroplasty
MeSH Terms: interventions — Gait Analysis; Biomechanical Phenomena; Kinetics

STUDY DESIGN:
Who Masked: Participant
Masking Description: Preop Postop
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative (Experimental): Gait analysis kinematics and kinetics
  Interventions: Other: Gait analysis
- Postoperative (Experimental): Gait analysis kinematics and kinetics
  Interventions: Other: Gait analysis

INTERVENTIONS:
Other: Gait analysis — Gait analysis
  Other Names: Kinematics and kinetics

SUMMARY:
The primary goal of Total Hip Replacement (THR) surgery in the treatment of hip osteoarthritis is to reduce pain and restore hip function in order to increase patient mobility and quality of life. Two different cement fixation methods are used in order to insert THR implants. This will be done before and after surgery in 2 groups randomized to either of 2 cement fixation methods. Gait analysis preoperative and 2 year after surgery.

DETAILED DESCRIPTION:
The primary goal of Total Hip Replacement (THR) surgery in the treatment of hip osteoarthritis is to reduce pain and restore hip function in order to increase patient mobility and quality of life. Patients with radiological signs of osteoarthritis of the hip, hip pain and functional disability may be treated with insertion of a THA.

Two different fixation methods are used in order to insert THR implants. Cemented fixation using bone cement, polymethyl methacrylate (PMMA) is the most commonly used fixation method in Sweden. A new bone cement, Refobacin®, already marketed in Germany is planned to be introduced in Sweden in late 2018.

The hospital is also equipped with a modern gait laboratory were the functional gait performance can be evaluated. This will be done before and after surgery in 2 groups randomized to either of 2 cement fixation methods. The subjects will undergo gait analysis befor and 2 year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* hip arthritis

Exclusion Criteria:

* no hip arthritis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Kinematics | Preop
  Hip angels in 3 planes
Kinematics | Postop 2 year
  Hip angels in 3 planes

CONTACTS AND LOCATIONS:
Overall Officials: Roland Zügner, Principal Investigator — Göteborg University
Locations (1):
- Roland Zügner, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Plan to make individual participant data (IPD) after publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication
Access Criteria: After publication